CLINICAL TRIAL: NCT02486887
Title: Monitoring Electronique à Distance Des Patients Insuffisants Cardiaques
Brief Title: Home Electronic Monitoring of Chronic Heart Failure
Acronym: MEDIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: AG2R La Mondiale (Other); IMRI (Unknown); AFPEC (Unknown); H2AD (Other); Pôle des Microtechniques de Besançon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P/2014/234
Record Dates: First submitted 2015-06-01; First posted 2015-07-01 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Chronic Heart Failure
Keywords: telemonitoring
MeSH Terms: interventions — Heart Rate; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- telemonitoring (Experimental): telemonitoring of weight, arterial pressure and heart rate at home with connection to a medical platform to monitor the evolution.
  Interventions: Device: telemonitoring of weight, pulse and blood pressure
- conventional follow-up (No Intervention): conventional follow-up

INTERVENTIONS:
Device: telemonitoring of weight, pulse and blood pressure
  Arms: telemonitoring

SUMMARY:
The main objective of the study is to evaluate the effect of telemonitoring on mortality and rehospitalization due to heart failure on patients with chronic heart failure which have follow an educational program compared to a conventional follow-up during 1 year.

The secondary objectives of the study are :

* Evaluate the cost of health
* Qualitatively evaluate telemonitoring on uses
* Evaluate quality of life

DETAILED DESCRIPTION:
prospective, monocentric, randomized open-labeled study.

1. - Data collected

   1. - during inclusion visit sex, age, full contact details, marital status, number of child, level of education, professional status weight, height, BMI, cardiac pulse, blood pressure, NYHA, consumption of tobacco and alcohol, concomitant treatments, medical history BNP, prealbumin Quality of life questionnaire (Minnesota), Depression questionnaire (HAD), autonomy questionnaire (IADL)
   2. - at 6 month weight, height, BMI, cardiac pulse, blood pressure, NYHA, consumption of tobacco and alcohol, concomitant treatments, medical history BNP, prealbumin Number of consultations, nurses care, number of hospitalization in emergency care unit, number of hospitalization due to acute heart failure, number of days of hospitalization, number of medical transports Quality of life questionnaire (Minnesota), Depression questionnaire (HAD), autonomy questionnaire (IADL)
   3. - at one year weight, height, BMI, cardiac pulse, blood pressure, NYHA, consumption of tobacco and alcohol, concomitant treatments, medical history BNP, prealbumin Number of consultations, nurses care, number of hospitalization in emergency care unit, number of hospitalization due to acute heart failure, number of days of hospitalization, number of medical transports Quality of life questionnaire (Minnesota), Depression questionnaire (HAD), autonomy questionnaire (IADL)
2. - Medico-economic evaluation The objective of this evaluation is to analyzed the efficiency of telemonitoring in patients with chronic heart failure.

   This evaluation has to be :
   * quantitative : directs modifications of cost and nature of health care follow-up or organization
   * qualitative : indirect impact on health care costs of situations or behavior
3. - study of uses "uses" is faculty of recognition, comprehension, use, appropriation and diversion of the telemonitoring by patients.

During the first phase, interviews to obtain qualitative vision of interactions between telemonitoring and ecosystems of players.

40 qualitative interviews during 2 hours of : 30 patients ; 24 users of telemonitoring and 6 non-users. 10 members of medical and paramedical staff The objectives of the second phase is to defined usage scenarios from previous assessments.

4.- Telemonitoring surveillance of weight, blood pressure and cardiac pulse, 3 times a week by the patient at home.

H2AD platform, general practitioner, cardiology unit, therapeutical education team had to manage alarms.

The devices (balance, blood pressure and pulse monitor) are related by GPRS to a medical platform. The platform receive every measure of weight, blood pressure and pulse. When weight, blood pressure or pulse increased or decreased, alarms are emitted and patients are contacted by a practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure, NYHA II, III or IV
* Patients with follow-up in therapeutic education program and who had finish the program in 2011, 2012, 2013, 2014, 2015, 2016, 2017
* Information given and informed consent given

Exclusion Criteria:

* vital emergencies
* Refusal of patient, cardiologist or general practitioner
* Person who is not able to communicate or answer the questions
* Patients with problems of understanding as such dure to those diseases : dementia, Alzheimer disease, or neurological sequelae of cerebral stroke
* Patients who do not speak french
* Patients under guardianship
* Patients with other diseases which alter quality of life
* Patients who participate to another clinical trial
* Person private of liberty by court decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Number of rehospitalizations due to acute heart failure and number of death due to heart failure | 1 year

SECONDARY OUTCOMES:
Number and cost of consultations, treatments, hospitalization, transport, care of nurses ... | 1 year
Qualitative interviews of patients and to all medical care services about uses and services rendered by the new device | 1 year
Interviews of patients and comptability of alarms of non-observance of weight, pulse and arterial pressure measure to evaluate acceptability and observance of telemonitoring device | 1 year
Scores on questionnaires of minnesota, EQ-5D and IADL to evaluate quality of life and autonomy | 1 year
Mean duration of stay during hospitalization | 1 year
Number of hospitalization in emergency care unit to measure efficacy of telemonitoring | 1 year
Number of alarm for increase of weight, hypo- or hypertension, bradycardia or tachycardia as a measure of efficacy of telemonitoring | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France